CLINICAL TRIAL: NCT04562233
Title: Breast Cancer and Resistance Exercise Program (B-REP): A Feasibility and Acceptability Trial
Brief Title: Breast Cancer and Resistance Exercise Program
Acronym: B-REP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, CINJRegulatory, Administrative, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2020002182; Pro2020002182 (Other: Rutgers IRB); 132012 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Resistance Training
Keywords: online; breast cancer; physical activity; breast neoplasm; resistance exercise; survivor
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants will engage in 12, weekly, supervised, exercise sessions using Zoom with the exercise trainer. Once a week, the exercise trainer and participant will each log on to Zoom from their locations to begin the supervised exercise session. The exercise trainer will record all sessions. Sessions will be 30 to 45 minutes long and be structured as follows: review of previous session and an opportunity to ask questions; 5-minute warm-up; 20- to 25-minute workout; 5- to10-minute cool down and reminder of next session and/or data collection time period. Supervised sessions will be scheduled once a week over the 12-week intervention. Participants will be expected to complete their resistance-based physical activity program for an additional 1-2 days a week as per the intervention schedule to meet as physical activity guidelines. The exercise trainer will track participant attendance. During the session, participants must have another person in the same location in case of an emergency.
  Interventions: Behavioral: Online-delivered physical activity intervention.
- Control Arm (Other): The attention control arm will include a printed, individualized resistance-based physical activity program.
  Participants randomized to the control arm will be given a printed or digital individualized, resistance-based physical activity program and told to aim to for three exercise sessions per week. Control participants will follow the same measurement schedule as intervention participants.
  Interventions: Behavioral: Printed, individualized resistance-based physical activity program.

INTERVENTIONS:
Behavioral: Online-delivered physical activity intervention. — Participants randomized to the intervention arm will engage in 12, weekly, supervised, exercise sessions using Zoom with the exercise trainer.
  Arms: Intervention arm
Behavioral: Printed, individualized resistance-based physical activity program. — Without the supervision of an exercise trainer, participants will be given a printed, individualized resistance-based physical activity program to complete over the course of 12 weeks.
  Arms: Control Arm

SUMMARY:
The goal of the study is to test the feasibility and acceptability of a supervised, online-delivered, individualized, physical activity program in a sample of post-active treatment breast cancer survivors. The proposed intervention will use a 2-arm randomized controlled trial study design to compare a 12-week resistance-based physical activity program to an attention control (i.e., printed individualized physical activity program) group on feasibility, acceptability and changes in strength as measured by 10 repetition maximum (10RM). Both groups will wear accelerometers. The main hypothesis is that participants randomized to the intervention arm will rate the online-delivered physical activity program as feasible and acceptable compared to attention control participants. The overall rationale is that delivering a physical activity intervention online may increase uptake of the intervention, which may lead to maintained physical activity behavior and associated health benefits. The primary outcomes are feasibility as measured by participant retention and acceptability as measured by adherence to physical activity program (recorded by physical activity log). Secondary outcomes include changes in strength as measured by 10RM, objectively measured physical activity levels as measured by the accelerometer, satisfaction, physical functioning and health-related quality of life. Additionally, a select number of participants will be invited for an interview to talk about their experiences in the program, motivation and barriers to exercise.

Interview description: Participants will complete one-on-one interviews with the PI or research staff over videoconferencing software (Rutgers Zoom). The interview will be 45 to 60 minutes in duration and audio recorded using the "record meeting" function. Prior to the interview, participants will consent to being audio recorded. The recording will be stored on Box (a HIPAA compliant cloud drive). A transcript of the audio will be generated using the "audio transcript" function on Rutgers Zoom and transcribed by a third party to ensure accuracy.

DETAILED DESCRIPTION:
The project will use a 2-arm randomized controlled trial study. The intervention will include a 12, weekly, supervised, online-delivered, individualized resistance-based exercise program. The attention control arm will include a printed, individualized resistance-based physical activity program. A total of 50 breast cancer survivors will be recruited from Rutgers Cancer Institute of New Jersey (CINJ) and randomized to one of two study arms. The intervention arm will test the feasibility and acceptability of the intervention compared to the control arm, which will receive a printed or digital copy of an individualized physical activity program. Participants from both arms will receive an accelerometer (ActiGraph GT3X+), resistance bands (TheraBand®), and additional free weights (if required). Outcome measures will be assessed at baseline (pre-intervention), Week 12 (post-intervention) and Week 24 (follow-up). Data collection will occur both in-person and online. Data will be both objective (10RM, functional strength, physical activity measured by accelerometers, physical function assessments, and attendance) and subjective (self-reported physical activity program adherence, satisfaction, physical activity levels, health-related quality of life, and exercise and barrier self-efficacy).

Additionally, participants will complete one-on-one interviews with the PI or research staff over videoconferencing software (Rutgers Zoom). The interview will be 45 to 60 minutes in duration and participants will be asked to discuss their experiences in the program.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years and older
2. self-identify as Black or African American or Afro-Latina/e
3. a confirmed diagnosed of breast cancer < 10 years prior to study start
4. does not have a concurrent cancer diagnosis
5. have completed active treatment > 6 months prior to study commencement (hormonal therapy is acceptable)
6. who are inactive, defined as engaging in < 30 minutes of moderate-to-vigorous physical activity per day for 3 days per week
7. are able to exercise safely as per physical activity safety screening questionnaire, Get Active Questionnaire
8. read and understand English

h) have regular access to an internet-connected device with a video camera.

Exclusion Criteria:

1. respiratory, joint, or cardiovascular problems precluding physical activity as per physical activity safety screening questionnaire
2. metastatic disease
3. planned elective surgery during the duration of the intervention and/or follow-up that would interfere with participation (e.g., breast reconstruction surgery)
4. does not have someone to supervise them while they exercised remotely.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Feasibility (participant retention) | 14 weeks including pre-intervention and post-intervention questionnaire completion
  Participant retention at assessment timepoints (attendance and completing assessments)
Acceptability (program adherence) | 12 weeks to complete the intervention
  Adherence to physical activity program/intervention (attendance and exercise logs)
Internet Evaluation and Utility Questionnaire | After the 12 week intervention and captured in follow-up questionnaire for intervention arm participants
  Satisfaction will be measured as participants' experience and perceptions of an internet intervention. Scale values: Not at all, slightly, somewhat, mostly & very. Higher scores are associated with a greater level of satisfaction.

SECONDARY OUTCOMES:
10 Repetition Maximum Test | During the baseline assessment, week 12 assessment and week 24 follow up assessment
  Changes in strength measured by 10RM assessment
Godin Leisure Time Exercise Questionnaire | During the baseline assessment, week 12 assessment and week 24 follow up assessment
  Self-report exercise frequency (times per week) and intensity (mild, moderate, and vigorous). Higher scores indicate that individuals are more active.
Accelerometer (ActiGraph) | Prior to intervention start and following the Week 12 and week 24 assessments
  Objective measure of total physical activity levels with intensity and duration (minutes). No scale.
Senior Fitness Test | During the baseline assessment, week 12 assessment and week 24 follow up assessment
  Functional assessments including senior fitness test, which includes the 6 minute walk test, chair sit to stand test and arm curl test. Scores are compared to age-matched, national averages.
Exercise Self-Efficacy Questionnaire | During the baseline assessment, week 12 assessment and week 24 follow up assessment
  Confidence to exercise over the next three months rated on a scale of 0% to 100% confidence. High scores indicate higher perceived confidence to exercise.
Barrier Self-Efficacy Questionnaire | During the baseline assessment, week 12 assessment and week 24 follow up assessment
  Confidence to overcome commonly-reported barriers rated on a scale of 0% to 100%. Higher scores indicated higher perceived confidence to overcome barriers.
Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | Completed at baseline assessment, after completion of the intervention at week 12 and at the week 24 follow up
  Scale measures physical wellbeing, social/family wellbeing, emotional wellbeing and functional wellbeing with items specifically for breast cancer (additional concerns). Scale - Not at all, a little bit, some-what, quite a bit, very much. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fong, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data that underlie results will be shared after de-identification for analysis purposes. Data sources include: 1) clinical and physical assessment data collected at the CINJ, 2) patient-reported questionnaire data collected through REDCap in a personal device or study-specific iPad, 3) observational data collected from recording one-on-one exercise sessions, and 4) Interview audio from zoom and transcribed interviews
  The final dataset will not contain any information that could identify individuals. Data will be shared using secure, Rutgers email between the PI and Co-Is.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available to investigators after one month of data collection and up to 3 years after completion of research activities per Rutgers (ORRA) guidelines.
Access Criteria: Prior approved investigators authorized to review the data will have access to individual participant data.

REFERENCES:
- [Background] Ritterband LM, Bailey ET, Thorndike FP, Lord HR, Farrell-Carnahan L, Baum LD. Initial evaluation of an Internet intervention to improve the sleep of cancer survivors with insomnia. Psychooncology. 2012 Jul;21(7):695-705. doi: 10.1002/pon.1969. Epub 2011 Apr 29. PMID 21538678
- [Background] Amireault S, Godin G, Lacombe J, Sabiston CM. The use of the Godin-Shephard Leisure-Time Physical Activity Questionnaire in oncology research: a systematic review. BMC Med Res Methodol. 2015 Aug 12;15:60. doi: 10.1186/s12874-015-0045-7. PMID 26264621
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] McAuley E. Self-efficacy and the maintenance of exercise participation in older adults. J Behav Med. 1993 Feb;16(1):103-13. doi: 10.1007/BF00844757. PMID 8433355
- [Background] Get Active Questionnaire. Ottawa, Canada: Canadian Society of Exercise Physiology, 2016.
- [Background] Hilgart M, Ritterband L, Baxter K, Alfano A, Ratliff C, Kinzie M, Cohn W, Whaley D, Lord H, Garber S. Development and perceived utility and impact of a skin care Internet intervention. Internet Interventions. 2014;1(3):149-57. doi: 10.1016/j.invent.2014.07.003; PMCID: PMC Journal - In Process.
- [Derived] Fong AJ, Llanos AAM, Hudson SV, Schmitz K, Lu SE, Phillips SM, Manne SL. Online-delivered resistance exercise intervention among racially diverse breast cancer survivors: Feasibility, acceptability, and exploratory outcomes of B-REP. Support Care Cancer. 2024 Aug 1;32(8):565. doi: 10.1007/s00520-024-08769-9. PMID 39090218

DOCUMENTS (1):
  • Informed Consent Form (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT04562233/ICF_002.pdf